CLINICAL TRIAL: NCT03972046
Title: Neoadjuvant Use of Talimogene Laherparepvec and BRAF/MEK Inhibitor for Advanced Nodal BRAF Mutant Melanoma: A Pilot Study
Brief Title: Neoadjuvant Use of Talimogene Laherparepvec and BRAF/MEK Inhibitor for Advanced Nodal BRAF Mutant Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal investigator leaving study site; no replacement PI will be sought
Sponsor: TriHealth Inc. (Other)
Collaborators: TriHealth Cancer Institute (Unknown); TriHealth Surgical Institute (Unknown); TriHealth Ultrasound Department (Unknown); Bethesda North TriHealth Hospital (Unknown); Good Samaritan TriHealth Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-086; 20177504 (Other Grant/Funding Number: Amgen Inc.)
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-02

CONDITIONS: Melanoma (Skin); Melanoma Stage IIIb-IVM1a; Metastasis Skin; Tumor Skin; BRAF Gene Mutation
Keywords: T-VEC; BRAF/MEK inhibition; Melanoma; Nodal metastasis; Neoadjuvant treatment; BRAF mutant
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — talimogene laherparepvec; dabrafenib; trametinib

STUDY DESIGN:
Intervention Model Description: Patients, aged 18+, seen at the TriHealth Cancer Institute and/or TriHealth Surgical Institute with a palpable regional melanoma metastasis at the time of initial presentation or with regional recurrence and tumors with a BRAF mutation will be considered for participation in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- T-Vec + BRAF/MEK (Experimental): Participants will begin taking the following 3 medications:
  BRAF Inhibitor dabrafenib 150 mg by mouth twice a day; MEK inhibitor trametinib 2 mg by mouth once a day; Talimogene laherparepvec (T-Vec) up to 4mL subcutaneous injection (Dose #1: 10^6 PFU/mL; Dose #2: 10^8 PFU/mL 21 (+3) days after first dose; Subsequent doses: 10^8 PFU/mL every 14 (+/-3) days).
  Dosing to continue for at least 3 months, or up to 6 months if no plateau in response.
  May stop earlier than 3 months at physician discretion depending on side effects and response.
  Ultrasound of tumor nodal basin(s) monthly.
  Labs every 4 weeks: CBC with differential, CMP, LDH CT of chest/abdomen/pelvis every 3 months.
  PET CT or brain MRI as needed at discretion of the investigator.
  Manual tumor measurement in office prior to each injection.
  Interventions: Drug: Talimogene laherparepvec (T-Vec); Drug: Dabrafenib (BRAF Inhibitor); Drug: Trametinib (MEK Inhibitor)

INTERVENTIONS:
Drug: Talimogene laherparepvec (T-Vec) — Talimogene laherparepvec (T-Vec) up to 4mL subcutaneous injection
Drug: Dabrafenib (BRAF Inhibitor) — Dabrafenib (BRAF Inhibitor) 150 mg by mouth twice a day
Drug: Trametinib (MEK Inhibitor) — Trametinib (MEK Inhibitor) 2 mg by mouth once a day

SUMMARY:
This study will investigate whether the use of talimogene laherparepvec (T-VEC) in combination with BRAF/MEK inhibitor will result in durable regional and distant recurrence free survival in the neoadjuvant setting for treatment of advanced nodal BRAF mutant melanoma.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, open-label, single-center interventional study looking at the response rate when using talimogene laherparepvec (T-VEC) in combination with BRAF/MEK inhibitor in neoadjuvant setting for treatment of advanced nodal BRAF mutant melanoma. For this pilot study, a sample size of 20 participants, over 18 years of age will be included.

ELIGIBILITY:
Inclusion

* Age ≥ 18
* Malignant melanoma Stage IIIb-IVM1a patients.
* Primary or recurrent disease.
* Cutaneous primary melanoma or unknown primary.
* Measurable disease as evidenced by:

  * At least one lesion measuring greater than or equal to 10 mm on CT, ultrasound, or physical exam
  * A conglomerate of superficial lesions measuring which in aggregate have a total diameter of 10 mm
* Injectable disease
* Palpable regional metastasis at the time of initial presentation or with regional recurrence
* Tumor(s) with BRAF mutation
* ECOG 0,1,2
* Life expectancy > 2 years in the opinion of the investigator
* Able to provide written informed consent
* Adequate organ function based on most recent labs (according to investigator discretion), defined as follows:

  * Hematological: Absolute neutrophil count ≥ 1500/mm3 (1.5x109/L); Platelet count ≥ 75,000/mm3 (7.5x109/L); Hemoglobin ≥ 8 g/dL (without need for hematopoietic growth factor or transfusion support)
  * Renal: Serum creatinine ≤ 1.5 x upper limit of normal (ULN), OR 24-hour creatinine clearance ≥ 60 mL/min for subject with creatinine levels > 1.5 x ULN. (Note: Creatinine clearance need not be determined if the baseline serum creatinine is ≤ 1.5 x ULN. . Creatinine clearance should be determined per institutional standard).
  * Hepatic: Serum bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for a subject with total bilirubin level > 1.5 x ULN; Aspartate aminotransferase (AST) ≤ 2.5 x ULN OR ≤ 5 x ULN, if liver metastases present and injection does not involve a visceral lesion; Alanine aminotransferase (ALT) ≤ 2.5 x ULN OR ≤ 5 x ULN, if liver metastases present and injection does not involve a visceral lesion
  * Coagulation: International normalization ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN, unless the subject is receiving anticoagulant therapy, in which case PT and partial thromboplastin time (PTT)/ activated PTT (aPTT) must be within therapeutic range of intended use of anticoagulants; PTT or aPTT ≤ 1.5 x ULN, unless the subject is receiving anticoagulant therapy as long as PT and PTT/aPTT is within therapeutic range of intended use of anticoagulants.
  * Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to enrollment. If urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Exclusion

* BRAF wild type tumor
* M1b and M1c disease
* Clinically active cerebral metastases, bony metastases, visceral metastases
* Mucosal or ocular primary disease
* Known active central nervous system (CNS) metastases. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids >10 mg/day of prednisone or equivalent. The exception does not include carcinomatosus meningitis which is excluded regardless of clinical stability.
* History or evidence of active autoimmune disease that requires systemic treatment (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Evidence of clinically significant immunosuppression such as the following:

  * Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease.
  * Concurrent opportunistic infection.
  * Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 7 days prior to enrollment.
* Active herpetic skin lesions or prior complications of HSV-1 infection (e.g., herpetic keratitis or encephalitis).
* Requires intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (e.g., acyclovir), other than intermittent topical use.
* Previous treatment with talimogene laherparepvec or any other oncolytic virus.
* Previous treatment with a BRAF or MEK inhibitor
* Prior therapy with tumor vaccine.
* Received live vaccine within 28 days prior to enrollment.
* Prior immunosuppressive, chemotherapy, radiotherapy (in which the field encompassed a planned injection site), biological cancer therapy, or major surgery within 28 days prior to enrollment or has not recovered to CTCAE grade 1 or better from adverse event due to cancer therapy administered more than 28 days prior to enrollment. Adjuvant hormonal therapy is allowed if appropriate for planned study.
* Prior radiotherapy in which the field does not overlap the injection sites or non-immunosuppressive targeted therapy within 14 days prior to enrollment or has not recovered to CTCAE grade 1 or better from adverse event due to cancer therapy administered more than 14 days prior to enrollment
* Currently receiving treatment with another investigational device or drug study, or < 28 days since ending treatment with another investigational device or drug study(s).
* Other investigational procedures while participating in this study are excluded.
* Known to have acute or chronic active hepatitis B infection.
* Known to have acute or chronic active hepatitis C infection.
* Known to have human immunodeficiency virus (HIV) infection.
* History of other malignancy within the past 5 years with the following exceptions:

  * Adequately treated non melanoma skin cancer without evidence of disease at the time of enrollment
  * Adequately treated cervical carcinoma in situ without evidence of disease at the time of enrollment
  * Adequately treated breast ductal carcinoma in situ without evidence of disease at the time of enrollment
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer at the time of enrollment.
* Subject has known sensitivity to talimogene laherparepvec or any of its components to be administered during dosing.
* Female subject is pregnant or breast-feeding, or planning to become pregnant during study treatment and through 3 months after the last dose of talimogene laherparepvec.
* Sexually active subjects and their partners unwilling to use male or female latex condom to avoid potential viral transmission during sexual contact while on treatment and within 30 days after treatment with talimogene laherparepvec.
* Subjects who are unwilling to minimize exposure with his/her blood or other body fluids to individuals who are at higher risks for HSV-1 induced complications such as immunosuppressed individuals, individuals known to have HIV infection, pregnant women, or infants under the age of 3 months, during talimogene laherparepvec treatment and through 30 days after the last dose of talimogene laherparepvec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Rate of recurrence-free survival | 1 year

SECONDARY OUTCOMES:
Rate of melanoma specific survival | 1 year
Rate of melanoma specific survival | 2 years
Rate of melanoma specific survival | 3 years
Rate of distant metastatic free survival | 1 year
Rate of distant metastatic free survival | 2 years
Rate of distant metastatic free survival | 3 years
Tumor response rate to therapy according to RECIST criteria | 3 months
Tumor response rate to therapy according to RECIST criteria | 6 months
Rate of pathological response in the surgical specimen | 3 months
Rate of pathological response in the surgical specimen | 6 months
Incidence of all adverse events (AEs) | 1 month
  includes treatment-related AEs, serious AEs, and fatal AEs
Incidence of all adverse events (AEs) | 2 months
  includes treatment-related AEs, serious AEs, and fatal AEs
Incidence of all adverse events (AEs) | 3 months
  includes treatment-related AEs, serious AEs, and fatal AEs
Incidence of all adverse events (AEs) | 4 months
  includes treatment-related AEs, serious AEs, and fatal AEs
Incidence of all adverse events (AEs) | 5 months
  includes treatment-related AEs, serious AEs, and fatal AEs
Incidence of all adverse events (AEs) | 6 months
  includes treatment-related AEs, serious AEs, and fatal AEs
Incidence of all adverse events (AEs) | 7 months
  includes treatment-related AEs, serious AEs, and fatal AEs

CONTACTS AND LOCATIONS:
Locations (1):
- TriHealth Cancer Institute - Kenwood, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flaherty KT, Infante JR, Daud A, Gonzalez R, Kefford RF, Sosman J, Hamid O, Schuchter L, Cebon J, Ibrahim N, Kudchadkar R, Burris HA 3rd, Falchook G, Algazi A, Lewis K, Long GV, Puzanov I, Lebowitz P, Singh A, Little S, Sun P, Allred A, Ouellet D, Kim KB, Patel K, Weber J. Combined BRAF and MEK inhibition in melanoma with BRAF V600 mutations. N Engl J Med. 2012 Nov 1;367(18):1694-703. doi: 10.1056/NEJMoa1210093. Epub 2012 Sep 29. PMID 23020132
- [Background] Andtbacka RH, Ross M, Puzanov I, Milhem M, Collichio F, Delman KA, Amatruda T, Zager JS, Cranmer L, Hsueh E, Chen L, Shilkrut M, Kaufman HL. Patterns of Clinical Response with Talimogene Laherparepvec (T-VEC) in Patients with Melanoma Treated in the OPTiM Phase III Clinical Trial. Ann Surg Oncol. 2016 Dec;23(13):4169-4177. doi: 10.1245/s10434-016-5286-0. Epub 2016 Jun 24. PMID 27342831
- [Background] Andtbacka RH, Kaufman HL, Collichio F, Amatruda T, Senzer N, Chesney J, Delman KA, Spitler LE, Puzanov I, Agarwala SS, Milhem M, Cranmer L, Curti B, Lewis K, Ross M, Guthrie T, Linette GP, Daniels GA, Harrington K, Middleton MR, Miller WH Jr, Zager JS, Ye Y, Yao B, Li A, Doleman S, VanderWalde A, Gansert J, Coffin RS. Talimogene Laherparepvec Improves Durable Response Rate in Patients With Advanced Melanoma. J Clin Oncol. 2015 Sep 1;33(25):2780-8. doi: 10.1200/JCO.2014.58.3377. Epub 2015 May 26. PMID 26014293
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Coit DG, Thompson JA, Algazi A, Andtbacka R, Bichakjian CK, Carson WE 3rd, Daniels GA, DiMaio D, Ernstoff M, Fields RC, Fleming MD, Gonzalez R, Guild V, Halpern AC, Hodi FS Jr, Joseph RW, Lange JR, Martini MC, Materin MA, Olszanski AJ, Ross MI, Salama AK, Skitzki J, Sosman J, Swetter SM, Tanabe KK, Torres-Roca JF, Trisal V, Urist MM, McMillian N, Engh A. Melanoma, Version 2.2016, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2016 Apr;14(4):450-73. doi: 10.6004/jnccn.2016.0051. PMID 27059193
- [Background] Thiam A, Zhao Z, Quinn C, Barber B. Years of life lost due to metastatic melanoma in 12 countries. J Med Econ. 2016;19(3):259-64. doi: 10.3111/13696998.2015.1115764. Epub 2015 Nov 25. PMID 26531249
- [Background] Solit DB, Rosen N. Resistance to BRAF inhibition in melanomas. N Engl J Med. 2011 Feb 24;364(8):772-4. doi: 10.1056/NEJMcibr1013704. No abstract available. PMID 21345109
- [Background] Hauschild A, Grob JJ, Demidov LV, Jouary T, Gutzmer R, Millward M, Rutkowski P, Blank CU, Miller WH Jr, Kaempgen E, Martin-Algarra S, Karaszewska B, Mauch C, Chiarion-Sileni V, Martin AM, Swann S, Haney P, Mirakhur B, Guckert ME, Goodman V, Chapman PB. Dabrafenib in BRAF-mutated metastatic melanoma: a multicentre, open-label, phase 3 randomised controlled trial. Lancet. 2012 Jul 28;380(9839):358-65. doi: 10.1016/S0140-6736(12)60868-X. Epub 2012 Jun 25. PMID 22735384
- [Background] Johnson AS, Crandall H, Dahlman K, Kelley MC. Preliminary results from a prospective trial of preoperative combined BRAF and MEK-targeted therapy in advanced BRAF mutation-positive melanoma. J Am Coll Surg. 2015 Apr;220(4):581-93.e1. doi: 10.1016/j.jamcollsurg.2014.12.057. Epub 2015 Jan 30. PMID 25797743
- [Background] Grigg C, Blake Z, Gartrell R, Sacher A, Taback B, Saenger Y. Talimogene laherparepvec (T-Vec) for the treatment of melanoma and other cancers. Semin Oncol. 2016 Dec;43(6):638-646. doi: 10.1053/j.seminoncol.2016.10.005. Epub 2016 Oct 27. PMID 28061981